CLINICAL TRIAL: NCT01159639
Title: Dual Antiplatelet Therapy in Patients With Aspirin Resistance Following Coronary Artery Bypass Grafting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zagreb (Other)
Responsible Party: Hrvoje Gasparovic,MD.PhD, Medical school, University of Zagreb, University hospital center Zagreb-Rebro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 8.1-10/41-2
Record Dates: First submitted 2010-07-08; First posted 2010-07-09 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2010-06

CONDITIONS: Coronary Artery Disease; Aspirin Resistance
Keywords: aspirin resistance; coronary artery bypass grafting; multiple electrode aggregometry; multiplate
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- aspirin low responders monotherapy (No Intervention): patients with inappropriate response to aspirin assessed by multiple electrode aggregometry
- aspirin low responders dual antiplatelet therapy (Active Comparator): patients with inappropriate response to aspirin 300 mg therapy after CABG, randomized to receive clopidogrel 75 mg in addition to aspirin
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — patients with inappropriate response to aspirin 300 mg after CABG, assessed by multiple electrode aggregometry are randomized to receive clopidogrel 75 mg daily dose
  Arms: aspirin low responders dual antiplatelet therapy

SUMMARY:
Reactive platelet hyperactivity following coronary artery bypass grafting (CABG) might lead to thrombotic complications and major ischemic cardiac events. The aim of this study is to evaluate the changes in platelet reactivity following CABG and to clarify a potentially beneficial effect of dual antiplatelet therapy in the group of patients with documented aspirin resistance following CABG. Platelet function will be assessed by multiple electrode aggregometry. Aortocoronary vein graft disease is comprised of three distinct but interrelated pathological processes: thrombosis, intimal hyperplasia and atherosclerosis. Early vein thrombosis is a major cause of vein graft attrition during the first month after CABG.

Bypass patency can be improved with antiplatelet therapy which is the mainstay of treatment for patients after CABG. A beneficial effect of acetylsalicylic acid (ASA) on vein graft patency has been previously shown. Some patients experience thrombotic events despite continuous aspirin administration after CABG. The investigators hypothesized that low responsiveness to aspirin might be a precipitating factor for adverse thrombotic events following CABG.

Low responsiveness to ASA, as assessed by platelet function tests, varies widely among patients. The etiology of postoperative platelet hyperactivity remains to be elucidated.

In this study a new point-of-care assay named multiple electrode aggregometry (MEA) using a device called Multiplate analyzer (Dynabyte, Munich, Germany) has been utilized. It allows for rapid and standardized assessment of platelet function parameters.

This is a prospective randomized trial. The aim of the study is to document whether introduction of dual antiplatelet therapy in patients with ASA resistance will lead to a lower incidence of major adverse cardiac events (MACE) at a six month follow up. The composite endpoint will include death, non-fatal myocardial infarction, stroke and cardiac rehospitalization. All patients will receive 300 mg of ASA starting 6 hours after surgery, provided that the chest tube output is minimal. On postoperative day 4 their platelet function will be assessed using the above mentioned MEA. The patients found to be aspirin resistant will then undergo the process of randomization. The first arm will include patients with ASA resistance in whom no additional antiaggregation will be administered. In the second arm the investigators will include patients who were randomized to receive 75 mg of clopidogrel in addition to the standard antiplatelet regimen of 300 mg of ASA.

Platelet function monitoring allows for individual tailoring of the antiplatelet therapy. The goal of this study is to define whether this strategy will lead to improved patient outcomes. Both major and minor bleeding complications will be strictly monitored and reported.

ELIGIBILITY:
Inclusion Criteria:

* Isolated coronary artery bypass grafting
* Patients older than 18 years
* Written informed consent
* Accurate antiplatelet therapy administration documentation

Exclusion Criteria:

* Missing consent
* Patients with cardiac surgical procedures other than isolated CABG
* Antiplatelet therapy other than aspirin 300 mg after CABG
* Previous PCI requiring clopidogrel therapy after CABG
* Patients with unknown preoperative anti-platelet status
* Urgent or emergent surgery
* Off-pump CABG
* Re-Do CABG
* Patients younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
MACE events | 6 months
  MACE: death; non-fatal myocardial infarction; stroke; cardiac rehospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Medical school Zagreb, University hospital center Zagreb, Zagreb, Croatia, Croatia

REFERENCES:
- [Derived] Kopjar T, Petricevic M, Gasparovic H, Svetina L, Milicic D, Biocina B. Postoperative Atrial Fibrillation Is Associated With High On-Aspirin Platelet Reactivity. Ann Thorac Surg. 2015 Nov;100(5):1704-11. doi: 10.1016/j.athoracsur.2015.05.001. Epub 2015 Jul 26. PMID 26215778
- [Derived] Petricevic M, Kopjar T, Gasparovic H, Milicic D, Svetina L, Zdilar B, Boban M, Mihaljevic MZ, Biocina B. Impact of aspirin resistance on outcomes among patients following coronary artery bypass grafting: exploratory analysis from randomized controlled trial (NCT01159639). J Thromb Thrombolysis. 2015 May;39(4):522-31. doi: 10.1007/s11239-014-1127-9. PMID 25095738
- [Derived] Gasparovic H, Petricevic M, Kopjar T, Djuric Z, Svetina L, Biocina B. Impact of dual antiplatelet therapy on outcomes among aspirin-resistant patients following coronary artery bypass grafting. Am J Cardiol. 2014 May 15;113(10):1660-7. doi: 10.1016/j.amjcard.2014.02.024. Epub 2014 Mar 1. PMID 24666617
- [Derived] Gasparovic H, Petricevic M, Kopjar T, Djuric Z, Svetina L, Biocina B. Dual antiplatelet therapy in patients with aspirin resistance following coronary artery bypass grafting: study protocol for a randomized controlled trial [NCT01159639]. Trials. 2012 Aug 25;13:148. doi: 10.1186/1745-6215-13-148. PMID 22920307